CLINICAL TRIAL: NCT04474925
Title: A Randomized Controlled Trial of Pre-operative Versus Post-operative Stereotactic Radiosurgery for Patients With Surgically Resectable Brain Metastases
Brief Title: Pre- Versus Post-operative SRS for Resectable Brain Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0010
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Brain Metastases
Keywords: Neurosurgery; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical Resection followed by SRS (Non-Experimental) (Active Comparator): Surgical Resection followed by SRS within 3 weeks of surgery date.
  Interventions: Procedure: Brain Surgery; Radiation: Stereotactic Radiosurgery
- SRS followed by Surgical Resection (Experimental) (Experimental): SRS followed by surgery within 1 week of radiotherapy end date.
  Interventions: Procedure: Brain Surgery; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Brain Surgery — Surgery to remove brain metastases
Radiation: Stereotactic Radiosurgery — SRS uses many focused radiation beams to treat tumors within the brain
  Other Names: SRS

SUMMARY:
The purpose of this study is to determine if performing radiotherapy (SRS) prior to surgery results in better treatment outcomes than performing surgery before radiotherapy for patients with brain metastases.

Brain metastases occur when cancer cells from a primary cancer (e.g. lung, breast, colon) travel through the bloodstream and spread (metastasize) to the brain. As these new tumors grow they apply pressure and change how healthy brain tissue works. This can lead to a loss of brain function and worsening quality of life. Treatments for patients whose cancer has spread to the brain is often surgery, radiation therapy (radiotherapy) or a combination of both.

Surgery is one the main treatments for brain tumors. To remove the tumor, a neurosurgeon makes an opening in the skull and attempts to the remove the entire tumor. If the tumor is too close to important brain tissue, the surgeon may attempt to remove part of the tumor. Removal of the tumor from the brain tissue is called resection. The complete or partial removal of tumor helps to relieve symptoms by reducing pressure on healthy tissues and reduces the amount of tumor that needs to be treated by radiotherapy.

One type of radiotherapy used to treat brain metastases is stereotactic radiosurgery (SRS). SRS uses many focused radiation beams to treat tumors within the brain. Unlike surgery, there is no incision or cut being made. Instead, SRS uses an accurate map of your brain to deliver a precise beam of radiation to the tumors. The radiation damages the tumor cells forcing them to shrink and die off. The focused radiation beams also limit damage to healthy brain tissue minimizing side effects.

Surgery followed by radiotherapy is a standard treatment for brain metastases. However, there are still risks associated with the combination of treatments. This study plans to investigate whether performing surgery prior to SRS results in improved quality of life and decreased side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pathologically-proven primary malignancy
* ECOG 0-2
* Ability to complete neurocognitive testing without assistance from family or friends.
* Previous SRS to lesions other than the one being resected is allowed
* Patients of childbearing / reproductive potential must have a negative urine or serum pregnancy test ≤7 days before enrollment
* Participants capable of giving informed consent, or if appropriate participants having an acceptable individual capable of giving consent

Exclusion Criteria:

* Patients who have received prior WBRT, or SRS to the lesion being resected at time of study accrual
* Patients unable to undergo MRI scan (e.g. pacemaker)
* Leptomeningeal disease
* Germ cell tumor, small cell lung cancer or hematological primary malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Local Control | This will be assessed at 12 months
  To compare local control (in months) of pre-operative versus post-operative SRS

SECONDARY OUTCOMES:
Local Control | This will be assessed at 6 and 24 months.
  To compare local control (in months) of pre-operative versus post-operative SRS
Distant Brain Recurrence Rate | This will be assessed at 6,12 and 24 months.
  To compare Distant Brain Recurrence Rate (%) of pre-operative versus post-operative SRS
Leptomeningeal Recurrence Rate | This will be assessed at 6,12 and 24 months.
  To compare the Leptomeningeal Recurrence Rate (%) of pre-operative versus post-operative SRS
Overall Survival | This will be assessed at 6,12 and 24 months.
  Overall survival will be compared between both treatment arms
Hopkins Verbal Learning Test | This will be assessed at 3,6,9,12,16 and 24 months.
  Participants are scored using a points based system on Total Recall, Delayed Recall, Retention (% retained), and a Recognition Discrimination Index.
Controlled Oral Word Association | This will be assessed at 3,6,9,12,16 and 24 months.
  Participants are scored on their ability to generate words starting with a specific letter in a one minute timeframe.
Trial Making Tests | This will be assessed at 3,6,9,12,16 and 24 months.
  Participants are scored on their ability to complete the test within a certain timeframe.

CONTACTS AND LOCATIONS:
Locations (1):
- Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das S, Faruqi S, Nordal R, Starreveld Y, Kelly J, Bowden G, Amanie J, Fairchild A, Lim G, Loewen S, Rowe L, Wallace C, Ghosh S, Patel S. A phase III, multicenter, randomized controlled trial of preoperative versus postoperative stereotactic radiosurgery for patients with surgically resectable brain metastases. BMC Cancer. 2022 Dec 30;22(1):1368. doi: 10.1186/s12885-022-10480-z. PMID 36585629